CLINICAL TRIAL: NCT02204345
Title: Open Label Phase Ib/II, Multicenter Study of the Combination of RO5479599 With Carboplatin and Paclitaxel in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) of Squamous Histology Who Have Not Received Prior Chemotherapy or Targeted Therapy for NSCLC
Brief Title: A Study Evaluating RO5479599 in Combination With Carboplatin and Paclitaxel in Participants With Advanced or Metastatic Non-Small-Cell Lung Cancer (NSCLC) of Squamous Histology
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP29360; 2014-001498-15 (EudraCT Number)
Record Dates: First submitted 2014-07-24; First posted 2014-07-30 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Carboplatin; Paclitaxel; lumretuzumab

ARMS (1):
- RO5479599 + Carboplatin + Paclitaxel (Experimental): RO5479599 800 milligrams (mg) will be administered in the Safety Run-In Phase by intravenous infusion q3w on Day 1 of 3-weekly cycles (each cycle of 21 days) in combination with carboplatin (to produce an area under the curve [AUC] of 6 mg/milliliter [mL]*minute) and paclitaxel 200 mg per square meter (mg/m^2) by intravenous infusion q3w for 4 to 6 cycles. Thereafter, RO5479599 will be continued as a monotherapy (carboplatin and paclitaxel may be continued at the investigator's discretion) until disease progression, death, unacceptable toxicity, withdrawal of consent, or study termination by sponsor, whichever occurs first.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: RO5479599

INTERVENTIONS:
Drug: Carboplatin — Carboplatin by intravenous infusion q3w for 4-6 cycles and thereafter as per investigator's discretion.
Drug: Paclitaxel — Paclitaxel by intravenous infusion q3w until disease progression, death, unacceptable toxicity or withdrawal of consent.
Drug: RO5479599 — RO5479599 will be administered as an intravenous infusion q3w until disease progression, death, unacceptable toxicity or withdrawal of consent.

SUMMARY:
A multi-center Phase Ib/II study of the combination of RO5479599 with carboplatin and paclitaxel once in every 3 week (q3w) regimen to evaluate the safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Locally advanced or metastatic (stage IIIB or IV) squamous NSCLC
* No prior systemic chemotherapy, targeted therapy for metastatic NSCLC
* Evidence of at least one radiologically measurable lesion as per RECIST version 1.1
* Adequate hematological, liver and renal function
* Participants must agree to either remain completely abstinent or to use effective contraceptive methods from screening until 6 months after the last dose of study treatment
* Histologically confirmed squamous NSCLC participants eligible for enrollment must provide archival tumor biopsy tissue or if unavailable must be willing to undergo a fresh pretreatment primary tumor or metastatic biopsy
* Participants with Gilbert's Syndrome will be eligible for the study

Exclusion Criteria:

* Concurrent therapy with any other investigational drug
* History or clinical evidence of central nervous system (CNS) primary tumors or metastases
* Evidence of significant, uncontrolled concomitant diseases, which could affect compliance with the protocol or interpretation of results, including uncontrolled diabetes mellitus and/or significant cardiovascular disease or uncontrolled infection
* Any other diseases, metabolic dysfunction, a physical examination finding or a clinical laboratory finding, giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* Major surgery or significant traumatic injury less than (<) 28 days prior to the first study treatment infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Pregnant or breast-feeding women
* History of other malignancies that could affect compliance with protocol or interpretation of results. Participants with malignancies diagnosed more than 5 years prior to study day one, adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer are generally eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Baseline up to Day 342
Percentage of Participants With Objective Response as Assessed by Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Baseline until disease progression, death, unacceptable toxicity, or withdrawal of consent, whichever occurred first (assessed every 6 weeks from baseline [Cycle 1 Day 1] [Cycle length = 21 days] up to Day 342)

SECONDARY OUTCOMES:
Progression-free Survival (PFS) as Assessed Using RECIST v1.1 | Baseline until disease progression, death, unacceptable toxicity, or withdrawal of consent, whichever occurred first (assessed every 6 weeks from baseline [Cycle 1 Day 1] [Cycle length = 21 days] up to Day 342)
Overall survival (OS) | Baseline until disease progression, death, unacceptable toxicity, or withdrawal of consent, whichever occurred first (assessed every 6 weeks from baseline [Cycle 1 Day 1] [Cycle length = 21 days] up to Day 342)
Percentage of Participants With Disease Control as Assessed by Investigator Using RECIST v1.1 | Baseline until disease progression, death, unacceptable toxicity, or withdrawal of consent, whichever occurred first (assessed every 6 weeks from baseline [Cycle 1 Day 1] [Cycle length = 21 days] up to Day 342)
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of RO5479599 | Pre-dose(Hour 0); at end of infusion (infusion duration=approximately 2 hours) on Day 1 of each cycle (cycle length= 21 days) up to end of treatment (EOT, Day 314); 3-6, 24, 72, 168, 264, 336, 432, 480 hours post-dose on Day 1 of Cycle 1,4; at Day 342
Maximum Observed Plasma Concentration (Cmax) of RO5479599 | Pre-dose (Hour 0) and at end of infusion (infusion duration=approximately 2 hours) on Day 1 of each cycle (cycle length= 21 days) up to EOT (Day 314); 3-6, 24, 72, 168, 264, 336, 432, 480 hours post-dose on Day 1 of Cycle 1,4; at Day 342
Trough Concentration (Ctrough) of RO5479599 | Pre-dose (Hour 0) on Day 1 of each cycle (cycle length = 21 days) up to EOT (Day 314)
Total Clearance (CL) of RO5479599 | Pre-dose (Hour 0) and at end of infusion (infusion duration=approximately 2 hours) on Day 1 of each cycle (cycle length= 21 days) up to EOT (Day 314); 3-6, 24, 72, 168, 264, 336, 432, 480 hours post-dose on Day 1 of Cycle 1,4; at Day 342
Volume of Distribution at Steady State (Vss) of RO5479599 | Pre-dose (Hour 0) and at end of infusion (infusion duration=approximately 2 hours) on Day 1 of each cycle (cycle length= 21 days) up to EOT (Day 314); 3-6, 24, 72, 168, 264, 336, 432, 480 hours post-dose on Day 1 of Cycle 1,4; at Day 342
Accumulation Ratio (Rac) of RO5479599 | Pre-dose(Hour 0); at end of infusion (infusion duration=approximately 2 hours) on Day 1 of each cycle (cycle length= 21 days) up to end of treatment (EOT, Day 314); 3-6, 24, 72, 168, 264, 336, 432, 480 hours post-dose on Day 1 of Cycle 1,4; at Day 342
Terminal Elimination Half-life (t 1/2) of RO5479599 | Pre-dose(Hour 0); at end of infusion (infusion duration=approximately 2 hours) on Day 1 of each cycle (cycle length= 21 days) up to end of treatment (EOT, Day 314); 3-6, 24, 72, 168, 264, 336, 432, 480 hours post-dose on Day 1 of Cycle 1,4; at Day 342
Concentration of RO5479599 at the Time of Tumor Progression (Cprog) | At tumor progression (any time between Baseline and Day 342)
Concentration of RO5479599 at the Time of Tumor Response (Complete Response or Partial Response) | At the time of tumor response (anytime between baseline and Day 342)
Concentration of RO5479599 at the Time of Toxicity | At the time of toxicity (anytime between baseline and Day 342)
Concentration of RO5479599 at the Time of Infusion-related Reactions (IRRs) or Hypersensitivity Reaction | At the time of IRRs or Hypersensitivity Reaction (anytime between baseline and Day 342)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Toronto, Ontario, Canada
- København Ø, Denmark
- Spain (3):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Valencia, Valencia